CLINICAL TRIAL: NCT02526316
Title: Pilot Study on Concurrent Cisplatin-based Chemotherapy Combined With Vaccination Therapy With the P16_37-63 Peptide in Patients With HPV- and p16INK4a-positive Cancer
Brief Title: Cisplatin-based Chemotherapy Combined With P16_37-63 Peptide Vaccination in Patients With HPV-positive Cancers
Acronym: VICORYX-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oryx GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICORYX-2
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: HPV-induced Cancers
Keywords: cervical cancer; vulvar cancer; vaginal cancer; penile cancer; anal cancer; head and neck cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Penile Neoplasms; Anus Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- P16_37-63 Vaccination (Other): Patients will receive P16_37-63 peptide (100 μg) combined with Montanide® ISA-51 VG subcutaneously once a week for four weeks, followed by a 4 week rest period (1 cycle). The vaccination is to be started one week before the initiation or continuation of the cisplatin-based chemotherapy.
  Interventions: Biological: P16_37-63 peptide combined with Montanide® ISA-51 VG; Biological: P16_37-63 peptide without Montanide® ISA-51 VG

INTERVENTIONS:
Biological: P16_37-63 peptide combined with Montanide® ISA-51 VG — Patients will receive P16_37-63 peptide (100 µg) combined with Montanide® ISA-51 VG vaccination subcutaneously once a week for four weeks, followed by a 4 week rest period
Biological: P16_37-63 peptide without Montanide® ISA-51 VG — Patients will receive 30 mcg P16_37-63 peptide injected intradermally for test on delayed-type hypersensitivity (DTH) reactions.

SUMMARY:
The study will include 10 patients with HPV-associated ano-genital cancer (cervical, vulvar, vaginal, penile, anal) or HPV-associated head and neck cancer, who are planned to receive a cisplatin-based chemotherapy (alternatively a carboplatin-based chemotherapy may be selected by investigators choice). Patients will receive P16_37-63 peptide (100 µg) combined with Montanide® ISA-51 VG subcutaneously once a week for four weeks, followed by a 4 week rest period (1 cycle). The vaccination is to be started one week before the initiation or continuation of the cisplatin-based chemotherapy. Concurrent radiation is allowed and should be documented. The vaccination schedule will be repeated up to a total of 3 cycles (= 6 months) or until progression or intolerable toxicity. If chemotherapy is withheld (e.g. for toxicity), vaccination treatment can be continued.

DETAILED DESCRIPTION:
10 patients with HPV- and p16INK4a-positive cervical, vulvar, vaginal, penile, anal or head and neck cancer will be enrolled. The p16INK4a-peptide (p16INK4a-37-63, 100 mcg) mixed with MONTANIDE ISA-51 VG (0.3 ml) will be administered subcutaneously once weekly for four weeks, followed by a 4-week rest period (1 cycle). This schedule will be repeated for a total of 3 cycles (= 6 months) or until tumor progression or intolerable toxicity is documented. The first application will be done one week before chemotherapy initiation or continuation. Concurrent radiation is allowed and should be documented. If chemotherapy is withhold for toxicity, vaccination treatment can be continued.

Patients will be seen at baseline/screening and at every visit for safety assessment until disease progression or discontinuation of trial therapy for other reasons. Immunological assessments will be made in all patients. The immunological assessment includes the delayed time hypersensitivity response (DTH) against the P16_37-63 peptide. Therefore in week 1, 9, 17 and 25, 30 mcg P16_37-63 peptide solution without MONTANIDE ISA-51 VG will be injected at a separate site from the vaccination site intradermally. Immunological responses are evaluated at baseline and after vaccination in weeks 9, 17 and 25 (ELISPOT) and in weeks 1, 3, 9, 11, 17, 19 and 25 (ELISA) and are compared to the antigen-specific immune response measured before vaccination (week 1). Radiological tumor assessment (CT, MRI) will be performed at baseline and then every 8 weeks (after every cycle). There will be a follow- up visit four weeks after the last vaccination for safety. Further follow-up regarding progression and death can be performed, e.g. via a phone call. Autoimmunity will be assessed every 8 weeks. Safety of the immunization will be analyzed as assessed by the number and severity of adverse events categorized according to CTC criteria

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, advanced HPV-positive cervical, vulvar, vaginal, penile, anal or head and neck cancer cancer
* HPV positivity as tested by HPV genotyping from paraffin embedded tumor tissue using Linear Array HPV Genotyping test from Roche Diagnostics Germany GmbH
* Diffuse expression of p16INK4a in the tumor as analyzed by immunohistochemistry on paraffin embedded tumor tissue using the CINtec p16INK4a histology kit
* Planned cisplatin-based chemotherapy with an expected duration of at least 2 months. A carboplatin-based therapy may be selected as an alternative by investigators choice
* Expected survival of at least 3 months
* Full recovery from prior surgery, chemotherapy or radiation therapy (except for alopecia, fatigue or neurotoxicity of grade 1 or 2
* ECOG performance status 0, 1 or 2
* The following laboratory results: Neutrophil count ≥ 1.5 x 109/L Lymphocyte count ≥ 0.5 x 109/L Platelet count ≥ 100 x 109/L Serum bilirubin < 2mg/dL
* Patient´s written informed consent for participation in the trial

Exclusion Criteria:

* Prior treatment with P16_37-63 peptide
* Clinically significant heart disease (NYHA Class III or IV)
* Other serious illnesses, e.g., serious infections requiring antibiotics or bleeding disorders
* History of immunodeficiency disease or autoimmune disease
* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available
* Known HBV, HCV or HIV positivity
* Immunotherapy within 4 weeks before study entry
* Concomitant treatment with steroids, antihistaminic drugs, or nonsteroidal anti-inflammatory drugs (unless used in low doses for prevention of an acute cardiovascular event or for pain control). Topical or inhalational steroids are permitted
* Participation in any other clinical trial involving another investigational agent within 4 weeks
* Pregnancy or lactation
* Women of childbearing potential who are not using a medically acceptable means of contraception. Appropriate contraception is defined as surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), and double-barrier methods (any double combination of: intrauterine device, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap)
* Psychiatric or addictive disorders that may compromise the ability to give informed consent
* Lack of availability of a patient for immunological and clinical follow-up assessment
* Brain metastases (symptomatic and non-symptomatic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Immune response against peptide P16_37-63 | week 1
  A positive immune response is defined as positive DTH response against peptide P16_37-63 and/or a humoral (ELISA for the detection of p16-specific IgG/IgM/IgA) and/or CD4 cellular (IFN gamma ELISpot for the detection of p16INK4a-specific T cells) immune response exceeding the assay specific cut-off values for a positive response against peptide P16_37-63
Immune response against peptide P16_37-63 | week 3
  A positive immune response is defined as positive DTH response against peptide P16_37-63 and/or a humoral (ELISA for the detection of p16-specific IgG/IgM/IgA) and/or CD4 cellular (IFN gamma ELISpot for the detection of p16INK4a-specific T cells) immune response exceeding the assay specific cut-off values for a positive response against peptide P16_37-63
Immune response against peptide P16_37-63 | week 9
  A positive immune response is defined as positive DTH response against peptide P16_37-63 and/or a humoral (ELISA for the detection of p16-specific IgG/IgM/IgA) and/or CD4 cellular (IFN gamma ELISpot for the detection of p16INK4a-specific T cells) immune response exceeding the assay specific cut-off values for a positive response against peptide P16_37-63
Immune response against peptide P16_37-63 | week 11
  A positive immune response is defined as positive DTH response against peptide P16_37-63 and/or a humoral (ELISA for the detection of p16-specific IgG/IgM/IgA) and/or CD4 cellular (IFN gamma ELISpot for the detection of p16INK4a-specific T cells) immune response exceeding the assay specific cut-off values for a positive response against peptide P16_37-63
Immune response against peptide P16_37-63 | week 17
  A positive immune response is defined as positive DTH response against peptide P16_37-63 and/or a humoral (ELISA for the detection of p16-specific IgG/IgM/IgA) and/or CD4 cellular (IFN gamma ELISpot for the detection of p16INK4a-specific T cells) immune response exceeding the assay specific cut-off values for a positive response against peptide P16_37-63
Immune response against peptide P16_37-63 | week 19
  A positive immune response is defined as positive DTH response against peptide P16_37-63 and/or a humoral (ELISA for the detection of p16-specific IgG/IgM/IgA) and/or CD4 cellular (IFN gamma ELISpot for the detection of p16INK4a-specific T cells) immune response exceeding the assay specific cut-off values for a positive response against peptide P16_37-63
Immune response against peptide P16_37-63 | week 25
  A positive immune response is defined as positive DTH response against peptide P16_37-63 and/or a humoral (ELISA for the detection of p16-specific IgG/IgM/IgA) and/or CD4 cellular (IFN gamma ELISpot for the detection of p16INK4a-specific T cells) immune response exceeding the assay specific cut-off values for a positive response against peptide P16_37-63

SECONDARY OUTCOMES:
Tumor response as assessed by CT or MRI scans according to RECIST | baseline, after every cycle up to 25 weeks
Case wise listing of progression-free survival | four weeks after last vaccination
Safety of the vaccine administration as assessed by the number and severity of adverse events categorized according to CTC criteria version 4.0. | up tp week 25, 4 weeks after last vaccination
Case wise listing of overall survival | four weeks after last vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Krankenhaus Nordwest, Frankfurt, Germany